CLINICAL TRIAL: NCT02097563
Title: Family-Focused Therapy for Youth With Early-Onset Bipolar or Psychotic Disorders
Acronym: FFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, David J. Miklowitz, Ph.D., Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5R33MH097007 (NIH)
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Mood Disorders; Psychotic Disorders
Keywords: Mood Disorders; Psychosis; Subthreshold; Bipolar Disorder
MeSH Terms: conditions — Mood Disorders; Psychotic Disorders; Bipolar Disorder | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Intensity Training (Experimental): High intensity training: clinician attends a 6-hr live workshop in family-focused treatment techniques, and then, after taking on a case, gets weekly technical consultation sessions (by telephone) in FFT from an expert after every session;
  Interventions: Behavioral: High Intensity Training
- Low Intensity Training (Active Comparator): Low Intensity Training: clinician completes online workshop in FFT and then, after taking on a case, gets telephone consultation sessions after every third session.
  Interventions: Behavioral: Low Intensity Training

INTERVENTIONS:
Behavioral: High Intensity Training — This is a training method involving a live workshop followed by high intensity technical consultation.
  Arms: High Intensity Training
Behavioral: Low Intensity Training — Clinicians complete an online workshop in family-focused therapy, followed by technical consultation sessions after every third session.
  Arms: Low Intensity Training

SUMMARY:
The present study aims to :

1. compare different approaches (high intensity vs. low intensity) to training community providers (those who routinely treat young patients with bipolar disorder, psychosis, or sub-threshold high-risk conditions) on the implementation of family-focused treatment (FFT);
2. assess the cost of FFT training and implementation support; and
3. determine whether these different forms of clinician training are associated with different outcomes over 1 year among patients with early-onset mood and psychotic disorders.

DETAILED DESCRIPTION:
Despite impressive results in laboratory settings, there has been a significant lag in the community adoption and sustainability of family interventions for early-onset mood and psychotic disorders. Our objective is to determine the optimal methods of training and monitoring the delivery of an evidence-based family-focused treatment (FFT) in community providers who treat young patients (ages 13-25) with bipolar disorder (BD), psychosis, or "high-risk" conditions. FFT is administered in 12 sessions of psychoeducation, communication training, and problem-solving skills training. There are six randomized controlled trials indicating that, among adults or adolescents with BD, bipolar spectrum, or psychosis-risk disorders, FFT and pharmacotherapy are associated with more rapid stabilization of symptoms, delayed recurrences, enhanced functioning, better medication adherence, and improvements in family interaction relative to comparison treatments over 1-2 years. Using a community partnered participatory approach, we will engage diverse stakeholders (clinicians, administrators, caregivers) at three community sites (Harbor-UCLA Medical Center, San Fernando Mental Health Center, Didi Hirsch Mental Health Center) that treat early-onset, lower socioeconomic status, urban, and racially and ethnically diverse bipolar and psychosis patients. We will partner with these 3 community sites to randomly assign 30 clinicians to low intensity (web-based training plus low intensity supervision) or high intensity training (live workshop and higher intensity supervision, i.e., weekly individual supervision with fidelity feedback). Clinicians will administer FFT to up to 120 patients (ages 13-25) with recent-onset mania, psychosis or high-risk conditions. We expect that 20 clinicians will complete the treatment with 80 patients. Dependent variables will be empirically-derived fidelity component scores over time as measured by supervisors and clinicians. We hypothesize that after training, clinicians in both the high and low intensity groups will attain minimum levels of fidelity required for certification in the four components. However, clinicians in high intensity training will sustain higher levels of fidelity across subsequent treatment cases, and will be more satisfied and more likely to adopt the FFT model. This study will facilitate the translation of an evidence-based intervention and identify effective treatment components to inform larger-scale dissemination of FFT in community settings.

ELIGIBILITY:
Inclusion Criteria:

For patient participants:

Youth (13-17 years of age) and young adults (18-25 years of age) with the following:

1. Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) diagnosis of bipolar disorder (BD) type I or II;
2. DSM-5 diagnosis of schizophrenia, schizophreniform disorder, or psychosis not otherwise specified [NOS];
3. DSM-5 diagnosis of bipolar disorder, not elsewhere classified (formerly bipolar NOS; see criteria below); or
4. Research classification of ultra high-risk for psychosis.
5. at least one parent or step-parent with whom the subject lives is willing to participate in family treatment sessions;
6. the potential patient and relative(s) participants are able and willing to give written informed assent/consent to participate in the study.

Inclusion criteria for family clinicians:

1. works at one of the participating agencies (Harbor/UCLA, San Fernando Mental Health Center, Didi Hirsch Mental Health Services)
2. provides mental health care for youth or young adults with (or at risk for) bipolar or psychotic disorders
3. are licensed (medical, psychologist, clinical social work, marriage and family therapy) mental health provider or are eligible to be a licensed mental health provider (social work / psychology intern or extern, psychiatry resident, psychiatry child and adolescent psychiatry fellow) in the State of California working under the direct supervision of a licensed mental health professional.

Exclusion Criteria for patients:

1. a DSM-5 diagnosis of autism or pervasive developmental disorder, by history or medical records;
2. evidence of mental retardation by history or medical records (IQ < 70);
3. diagnosable and active substance or alcohol abuse or dependence disorders in the 4 months prior to study recruitment, although a lifetime history of substance or alcohol disorders can be present if the patient has been abstinent for at least 4 months;
4. a life-threatening medical disorder that requires immediate hospitalization or other emergency treatment;
5. evidence of current sexual or physical abuse of the child, and/or current domestic abuse between the adult partners. These situations usually require notification of the Department of Child Services and forms of treatment other than family therapy.

Exclusion criteria for clinicians: none.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Therapist Competency and Adherence Rating | One year
  This is a measure of how well the clinician administered family-focused treatment (FFT) based on ratings of audiotapes of family intervention sessions. These ratings are made every third session in both training conditions. This is an overall rating that can vary from 1 (nonadherent) to 7 (excellent adherence)

SECONDARY OUTCOMES:
Patient Health Questionnaire, 9 | 1 year
  Self-rating of depression and impairment, administered at baseline, 4 months, and 12 months
Young Mania Rating Scale | 1 year
  Mania symptoms (based on observer report) at baseline, 4 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David J Miklowitz, Ph.D., Principal Investigator — UCLA Semel Institute; Bowen Chung, M.D., Study Director — Harbor/UCLA Outpatient Psychiatry Program; Ira Lesser, M.D., Study Director — Harbor/UCLA Outpatient Psychiatry Program
Locations (3):
- United States (3):
  - Didi Hirsch Mental Health Services, Culver City, California
  - San Fernando Mental Health Center, Granada Hills, California
  - Harbor/UCLA Outpatient Psychiatry Porgram, Torrance, California

REFERENCES:
- [Background] Miklowitz DJ, Schneck CD, Singh MK, Taylor DO, George EL, Cosgrove VE, Howe ME, Dickinson LM, Garber J, Chang KD. Early intervention for symptomatic youth at risk for bipolar disorder: a randomized trial of family-focused therapy. J Am Acad Child Adolesc Psychiatry. 2013 Feb;52(2):121-31. doi: 10.1016/j.jaac.2012.10.007. Epub 2013 Jan 2. PMID 23357439
- [Derived] Miklowitz DJ, Weintraub MJ, Posta F, Denenny DM, Chung B. Effects of High- versus Low-Intensity Clinician Training on Implementation of Family-Focused Therapy for Youth with Mood and Psychotic Disorders. Fam Process. 2021 Sep;60(3):727-740. doi: 10.1111/famp.12646. Epub 2021 Mar 29. PMID 33779991
- See also: UCLA Child and Adolescent Mood Disorders Program — http://www.semel.ucla.edu/champ